CLINICAL TRIAL: NCT06350968
Title: Implementation of Online Advance Care Planning Tool for (Hemato-)Oncological Patients Within the Cancer Network Concord
Acronym: INDEED
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Maasstad Hospital (Other); Spijkenisse Medical Center (Unknown); Franciscus &Vlietland (Other); IJsselland (Unknown); Ikazia Hospital, Rotterdam (Other); Van Weel-Bethesda hospital (Unknown); Albert Schweitzer Hospital (Other); Beatrix hospital (Unknown)
Responsible Party: Principal Investigator, Wendy Oldenmenger, RN PhD, Principal Investigator, Erasmus Medical Center
Other Study IDs: MEC-2023-0151; 10200012110003 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2023-12-06; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Oncology; Advance Care Planning; Implementation
Keywords: Advance Care Planning; Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this mixed-methods study is to describe both the implementation process and outcomes of the online module Advance Care Plan for (hemato-)oncology patients within the oncology-network CONCORD.

The main question is: How is implementation and assurance of the advance care plan in daily care for (hemato-)oncological patients within CONCORD achieved, so that early integration of advance care planning in oncological care takes place and patient preferences are discussed?

Healthcare providers and patients are asked to use the module and share their experiences with it.

DETAILED DESCRIPTION:
Design Implementation research with a mixed-method design. Population

The implementation of advance care planning should benefit the care of (hemato-)oncology patients aged 18 years and older during the palliative phase of their illness. The research focuses on:

* Oncology patients who have been treated in one or more hospitals from the oncology-network CONCORD after their death (quantitative research)
* Oncology patients treated with palliative intent in one or more hospitals from this network (interviews)
* Healthcare providers and implementation staff in the relevant hospitals and from the service area (interviews) Goal The aim of this project is to implement advance care planning in (hemato-)oncology patients treated in one of the hospitals within the oncology-network CONCORD , so that personal preferences and treatment agreements lead to an appropriate treatment plan. This is examined through the process of implementation and assurance of advance care planning in oncological care.

MAIN QUESTION: How is implementation and assurance of the online module advance care planning in daily care for (hemato-)oncological patients within the oncology-network CONCORD achieved, so that early integration of advance care planning in oncological care takes place and patient preferences are discussed? Method

Qualitative research:

Description of the initial situation and the context within each institution, but also of general practitioners and patients using the NASSS Framework. Interviews with project leader, project coordinators in each hospital, healthcare providers from 1st, 2nd and 3rd lines, patients and relatives at the start and end of the project (3-5 in each target group per hospital, taking into account the greatest possible degree of diversity in age, gender and background). At the end of the project, the interviews are repeated to gather information about the experiences and lessons learned and the experiences with facilitating and hindering factors. Each interview is transcribed and analyzed using NVivio or Atlas.ti, analysis programs for qualitative data.

Quantitative research:

EHR-research based on anonymized data using a dashboard. A dashboard is being built in each hospital to analyze data from (hemato-)oncological patients who have been treated in the relevant hospital and have died. The dashboard contains demographic and medical data, the use of the proactive care module and medical consumption in the last three months of their lives.

In each of the participating hospitals, the (hemato-)oncological patients who died in the last 3 months of 2022, 2023, 2024 and 2025 are selected and it will be examined to what extent the advance care plan has been completed and what kind of care the patients have received. A 'Health economic analysis' is carried out using the data from the dashboard. On the one hand, this involves the costs of implementing the advance care planning module used. In addition, the dashboard maps medical consumption in the last three months of life (e.g. ICU admissions, ER visits, clinical admissions, etc.). This is translated into the nationally determined costs for this. This is done both before and after implementation has been mapped out among people who have died, making it possible to gain insight into the difference in costs incurred.

ELIGIBILITY:
Inclusion Criteria:

* Cancer
* Treated by hospital from the CONCORD-network

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with all types of (advanced)cancer.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Implementation outcome | 3 years
  Fidelity to the tailored implementation of the ACP-tool

SECONDARY OUTCOMES:
Intervention outcome | 3 years
  Healthcare use of patients with cancer in last phase of life (number of hospital admissions, ICU admissions, medication use, etc.)
Implementation outcome | 3 years
  Number of filled-in ACP-tools in EHR

CONTACTS AND LOCATIONS:
Locations (1):
- Joica Benschop, Rotterdam, Netherlands